CLINICAL TRIAL: NCT07056855
Title: Comparative Evaluation of Nano Hydroxy Apatite Varnish and Potassium Nitrate Gel Versus Fluoride Varnish as Non-invasive Treatment of Dentin Hypersensitivity in Permanent Teeth With Molar Incisor Hypo-mineralization: Randomized Clinical Trial
Brief Title: Three Different Topically Applied Materials as Non-invasive Treatment of Sensitivity in Permanent Teeth With Molar Incisor Hypomineralization
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mennat Allah Ashraf Abd Elsabour Abd Elkareem, Assistant Lecturer, Pediatric Dentistry Department, Ahram Canadian University. PhD student, Pediatric Dentistry and Dental Public Health Department, Cairo University. Affiliation: Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1444
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-03

CONDITIONS: Dentine Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessment of outcomes will be performed with two investigators other than the main investigator, who will not be aware of the type of the intervention carried out on the assessed child.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 8.6% nano-hydroxy apatite crystals varnish (Fygg's professional strength, Fygg, USA). (Experimental): Intervention group (1)
  Interventions: Drug: nano hydroxy apatite varnish Intervention (1)
- Potassium Nitrate (Ultradent UltraEZ Desensitizing Gel, Ultradent Inc., USA). (Experimental): Intervention group (2)
  Interventions: Drug: Potassium Nitrate Gel
- 5% fluoride varnish Control group (Active Comparator)
  Interventions: Drug: Varnishes, Fluorid

INTERVENTIONS:
Drug: nano hydroxy apatite varnish Intervention (1) — Fygg's professional strength, Fygg, USA
  Arms: 8.6% nano-hydroxy apatite crystals varnish (Fygg's professional strength, Fygg, USA).
Drug: Potassium Nitrate Gel — Ultradent UltraEZ Desensitizing Gel, Ultradent Inc., USA
  Arms: Potassium Nitrate (Ultradent UltraEZ Desensitizing Gel, Ultradent Inc., USA).
Drug: Varnishes, Fluorid — DentKist Charm Varnish 5% Sodium Fluoride Varnish
  Arms: 5% fluoride varnish Control group

SUMMARY:
This clinical study main goal is to investigate the effectiveness of nano hydroxy apatite crystal varnish and potassium nitrate gel as a non invasive approach in managing Dentin Hypersensitivity in MIH-affected teeth.

DETAILED DESCRIPTION:
This randomized clinical trial study aims to investigate the effectiveness of nano-hydroxy apatite crystal varnish, and potassium nitrate gel compared to fluoride varnish, in reducing dentin hypersensitivity, improving a child's oral hygiene.

ELIGIBILITY:
Participants related criteria:

1. Children aged from six to ten years old.
2. Medically free children according to the history taken from their parents.
3. Children who are categorized as Class I or II according to the American Society of Anaesthesiologists (ASA).
4. Children whom their parents accept to comply with the follow-up visits.
5. Children who accept, and their guardians, to participate in the study by signing the informed consent.

Tooth related criteria:

1. The diagnosis of MIH will be done as per the Wurzburg concept, 2023 MIH diagnostic criteria: The child will be confirmed to have MIH if any of the following characteristics are apparent:

* affected teeth show a clearly defined opacity at the occlusal and buccal surfaces of a tooth,
* defects vary in shape, size, and pattern,
* white, cream-colored, or yellow-brown color deviations are recognizable,
* defects variably vary in size,
* teeth with hypersensitivity are present,
* teeth have an atypical restoration,
* permanent teeth for (suspected) MIH reasons are missing (extractions),
* combinations of the above characteristics are present.

  1. MIH-affected permanent teeth, suffering from dentin hypersensitivity, (MIH-TNI 3).
  2. Positive Schiff Cold Airblasting Sensitivity score (score 1, 2, or 3).
* Exclusion criteria:

Participants related criteria:

1. Children with severe behavioral or emotional disabilities.
2. Children who received analgesics within the last 24 hours before the procedure.
3. Patients who are using chlorhexidine-based gels or mouthwashes.

Tooth related criteria:

1. A tooth with signs and symptoms of irreversible pulpitis.
2. A tooth with signs and symptoms of necrotic pulp.
3. Sealing therapy or application of desensitizing agent on the MIH teeth within one month before participation in the study.
4. Presence of dental caries on the MIH-affected permanent tooth.
5. Presence of restoration(s) on MIH-affected permanent tooth.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
Dentin Hypersensitivity | Baseline, 15 miutes pot-op, 2 weeks post-op, and 4 weeks post op
  Face scale: scores from 0-4. the higher the score the worse the sensitivity
Dentin Hypersensitivity | Baseline, 15 miutes pot-op, 2 weeks post-op, and 4 weeks post op
  chiff Cold Air Blasting Sensitivity Scale: scores from 0-3. The higher the score the worse the sensitivity.

SECONDARY OUTCOMES:
Oral hygiene | baseline, 2-, and 4- week post-op
  Measured by Plaque Control Record: Percentage.

IPD SHARING:
Plan to Share IPD: Undecided